CLINICAL TRIAL: NCT02469766
Title: A Comparison Between Flexible Ureteroscopy, Semirigid Ureteroscopy and Extracorporeal Shockwaves Lithotripsy (SWL) in The Management of Proximal Ureteric Stones. A Randomized Controlled Trial
Brief Title: Treatment of Upper Ureteric Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, muhamad muhamad abdallateef, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: upper ureteric stones
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Ureteric Stones
Keywords: ureteral stones; ureter; ureteroscopy; flexible; SWL

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extracorporeal Shockwaves (Active Comparator): Patients in this arm will undergo SWL
  Interventions: Procedure: SWL
- Semirigid URS (Active Comparator): Patients in this arm will undergo Semirigid Ureteroscopy
  Interventions: Procedure: Semirigid URS
- Flexible URS (Active Comparator): Patients in this arm will undergo Flexible Ureteroscopy
  Interventions: Procedure: Flexible URS

INTERVENTIONS:
Procedure: SWL — Patients in this arm will undergo SWL
  Arms: Extracorporeal Shockwaves
Procedure: Semirigid URS — Patients in this arm will undergo semirigid URS
  Arms: Semirigid URS
Procedure: Flexible URS — Patients in this arm will undergo Flexible URS
  Arms: Flexible URS

SUMMARY:
This study will be conducted to compare the success and complication rates of ureteroscopy, and shockwaves lithotripsy for treatment of upper ureteric stones ≤1 cm.

DETAILED DESCRIPTION:
This study will be conducted to compare the success and complication rates of Flexible, Semi-rigid URS, and SWL approaches for proximal ureteric stones with size ≤1 cm.

ELIGIBILITY:
Inclusion Criteria:

* Radio-opaque stones
* less than or equal 1 cm

Exclusion Criteria:

* Active UTI
* Coagulopathy
* Pregnancy
* Ureteric stricture

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 3 months
  The stone free rate will be evaluated with non-contrast CT

SECONDARY OUTCOMES:
Complication rate | 2 weeks
  Complications will be classified according to modified Clavien Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shoma, MD, Study Chair — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided